CLINICAL TRIAL: NCT05221866
Title: Efficiency And Quality In Post-Surgical Pain Therapy After Discharge
Acronym: EQUIPPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 0724-21-FB
Record Dates: First submitted 2021-10-26; First posted 2022-02-03 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Opioid Use; Opioid Dependence; Opioid Misuse; Post-Surgical Complication
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: The participant-facing app will be trialed prior to and after implementation of a provider-facing prescription intervention using a 2x2 design. Four arms will be described: the UControlPain App with Only data collection, the UControlPain Educational app only, the UControlPain App and provider-facing tool, and the UControlPain App with only data collection function and provider-facing tool. Once half of the subjects are enrolled, the provider-facing tool will be turned on.
Who Masked: Investigator
Masking Description: Randomization to the participant facing app will be implemented via REDCap. There will be no randomization in regard to the provider-facing intervention.The provider-facing intervention will be turned on once half the subjects are enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- UControlPain App With Only Data Collection Function (Control) (No Intervention): UControlPain App with only data collection function. No provider-facing prescription intervention.
- UControlPain Educational App Only (Active Comparator): UControlPain app with education components. No provider-facing prescription intervention.
  Interventions: Behavioral: Empowering Patient to Steer Their Pain Management After Surgery
- UControlPain App and Provider Facing Tool (Active Comparator): UControlPain app with education components and provider-facing prescription intervention. Once half of the subjects are enrolled, the provider-facing tool will be turned on. Participants will be masked to when the provider-facing tool is activated.
  Interventions: Behavioral: Empowering Patient to Steer Their Pain Management After Surgery; Behavioral: Provider-facing Prescription Aid
- Provider Facing Tool Only (Active Comparator): UControlPain App with only data collection function. Provider-facing prescription intervention. Once half of the subjects are enrolled, the provider-facing tool will be turned on. Participants will be masked to when the provider-facing tool is activated.
  Interventions: Behavioral: Provider-facing Prescription Aid

INTERVENTIONS:
Behavioral: Empowering Patient to Steer Their Pain Management After Surgery — Participants will be randomized to receive the consumer health informatics app (UControlPain) versus an app with only data collection function (no educational components) in an intent-to-treat design. Randomization will be implemented via REDCap by the study coordinators so that all investigators will remain blind to group assignment. Further, information on which type of app was installed will not be shared with providers or participants.
  Arms: UControlPain App and Provider Facing Tool; UControlPain Educational App Only
Behavioral: Provider-facing Prescription Aid — Providers will be given information to inform a participant-centered post-discharge pain management plan. This tool will be activated once half the subjects are enrolled. Participants will be masked when the provider-facing tool is turned on.
  Arms: Provider Facing Tool Only; UControlPain App and Provider Facing Tool

SUMMARY:
Following inpatient surgery, more than 80% of patients are prescribed opioids for use after discharge, yet up to 90% of patients report leftover opioids, and only 16% maximize non-opioid therapy. The proposed study seeks to test a provider-facing decision support tool and a participant-facing smartphone app to reduce the amount of opioids prescribed and taken following discharge, while ensuring effective treatment of pain after surgery. Adult participants with smart phones having had inpatient surgery requiring at least over-night hospitalization with anticipated discharge to home will be randomized to one of the two groups. Study measurements will include self-reported cumulative amounts of opioids taken after discharge, non-opioid analgesic taken, prescribed post-discharge opioid doses in morphine milligram equivalents (MME), pain intensity and pain interference scores (PROMIS), need for additional opioid prescriptions within one-month post-discharge, as well as any self-reported disposal of leftover medications.

DETAILED DESCRIPTION:
Prior to discharge from the hospital, patients will be approached regarding interest in the study with an introductory letter that describes the content and purpose of the study. Following informed consent, participants will be randomized to receive the consumer health informatics app (UControlPain) versus provision of an app with only data collection function (no educational components). Randomization will be implemented via REDCap by the study coordinators. Further, information on which type of app was installed will not be shared with providers or participants.

During the second half of the trial, a provider-facing electronic decision support tool will be activated. This will create a 2:2 design to test the provider-facing tool. Four arms will be described: the UControlPain App with Only data collection, the UControlPain Educational app only, the UControlPain App and provider-facing tool, and the UControlPain App with only data collection function and provider-facing tool. Once half of the subjects are enrolled, the provider-facing tool will be turned on.

ELIGIBILITY:
Inclusion Criteria:

* 19-89 years old
* Access to a smartphone (iOS or Android)
* Inpatient surgery requiring at least over-night hospitalization and anticipated discharge to home

Exclusion Criteria:

* Re-hospitalization within 30 days
* Pregnant
* Unable to read the English language
* Discharge to a post-acute care facility
* Contraindications to opioids, acetaminophen, or NSAIDs
* Long-term opioid therapy (AHRQ definition - opioid use on most days >3 months) prior to surgery

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Bartels, MD, PhD, MBA, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guy GP Jr, Zhang K, Bohm MK, Losby J, Lewis B, Young R, Murphy LB, Dowell D. Vital Signs: Changes in Opioid Prescribing in the United States, 2006-2015. MMWR Morb Mortal Wkly Rep. 2017 Jul 7;66(26):697-704. doi: 10.15585/mmwr.mm6626a4. PMID 28683056
- [Background] Scholl L, Seth P, Kariisa M, Wilson N, Baldwin G. Drug and Opioid-Involved Overdose Deaths - United States, 2013-2017. MMWR Morb Mortal Wkly Rep. 2018 Jan 4;67(5152):1419-1427. doi: 10.15585/mmwr.mm675152e1. PMID 30605448
- [Background] Bicket MC, Long JJ, Pronovost PJ, Alexander GC, Wu CL. Prescription Opioid Analgesics Commonly Unused After Surgery: A Systematic Review. JAMA Surg. 2017 Nov 1;152(11):1066-1071. doi: 10.1001/jamasurg.2017.0831. PMID 28768328
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Bateman BT, Cole NM, Maeda A, Burns SM, Houle TT, Huybrechts KF, Clancy CR, Hopp SB, Ecker JL, Ende H, Grewe K, Raposo Corradini B, Schoenfeld RE, Sankar K, Day LJ, Harris L, Booth JL, Flood P, Bauer ME, Tsen LC, Landau R, Leffert LR. Patterns of Opioid Prescription and Use After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):29-35. doi: 10.1097/AOG.0000000000002093. PMID 28594763
- [Background] Nooromid MJ, Blay E Jr, Holl JL, Bilimoria KY, Johnson JK, Eskandari MK, Stulberg JJ. Discharge prescription patterns of opioid and nonopioid analgesics after common surgical procedures. Pain Rep. 2018 Feb 6;3(1):e637. doi: 10.1097/PR9.0000000000000637. eCollection 2018 Jan. PMID 29430565
- [Background] Waljee JF, Li L, Brummett CM, Englesbe MJ. Iatrogenic Opioid Dependence in the United States: Are Surgeons the Gatekeepers? Ann Surg. 2017 Apr;265(4):728-730. doi: 10.1097/SLA.0000000000001904. No abstract available. PMID 27429023
- [Background] Howard R, Waljee J, Brummett C, Englesbe M, Lee J. Reduction in Opioid Prescribing Through Evidence-Based Prescribing Guidelines. JAMA Surg. 2018 Mar 1;153(3):285-287. doi: 10.1001/jamasurg.2017.4436. PMID 29214318
- [Background] Khorfan R, Shallcross ML, Yu B, Sanchez N, Parilla S, Coughlin JM, Johnson JK, Bilimoria KY, Stulberg JJ. Preoperative patient education and patient preparedness are associated with less postoperative use of opioids. Surgery. 2020 May;167(5):852-858. doi: 10.1016/j.surg.2020.01.002. Epub 2020 Feb 20. PMID 32087946
- [Background] Prabhu M, McQuaid-Hanson E, Hopp S, Burns SM, Leffert LR, Landau R, Lauffenburger JC, Choudhry NK, Kaimal A, Bateman BT. A Shared Decision-Making Intervention to Guide Opioid Prescribing After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):42-46. doi: 10.1097/AOG.0000000000002094. PMID 28594762
- [Background] Frieden TR, Houry D. Reducing the Risks of Relief--The CDC Opioid-Prescribing Guideline. N Engl J Med. 2016 Apr 21;374(16):1501-4. doi: 10.1056/NEJMp1515917. Epub 2016 Mar 15. No abstract available. PMID 26977701
- [Background] Manchikanti L, Helm S 2nd, Fellows B, Janata JW, Pampati V, Grider JS, Boswell MV. Opioid epidemic in the United States. Pain Physician. 2012 Jul;15(3 Suppl):ES9-38. PMID 22786464
- [Background] Heyward J, Olson L, Sharfstein JM, Stuart EA, Lurie P, Alexander GC. Evaluation of the Extended-Release/Long-Acting Opioid Prescribing Risk Evaluation and Mitigation Strategy Program by the US Food and Drug Administration: A Review. JAMA Intern Med. 2020 Feb 1;180(2):301-309. doi: 10.1001/jamainternmed.2019.5459. PMID 31886822
- [Background] Chen EY, Marcantonio A, Tornetta P 3rd. Correlation Between 24-Hour Predischarge Opioid Use and Amount of Opioids Prescribed at Hospital Discharge. JAMA Surg. 2018 Feb 21;153(2):e174859. doi: 10.1001/jamasurg.2017.4859. Epub 2018 Feb 21. PMID 29238810
- [Background] Carrico JA, Mahoney K, Raymond KM, McWilliams SK, Mayes LM, Mikulich-Gilbertson SK, Bartels K. Predicting Opioid Use Following Discharge After Cesarean Delivery. Ann Fam Med. 2020 Mar;18(2):118-126. doi: 10.1370/afm.2493. PMID 32152015
- [Background] Bartels K, Mahoney K, Raymond KM, McWilliams SK, Fernandez-Bustamante A, Schulick R, Hopfer CJ, Mikulich-Gilbertson SK. Opioid and non-opioid utilization at home following gastrointestinal procedures: a prospective cohort study. Surg Endosc. 2020 Jan;34(1):304-311. doi: 10.1007/s00464-019-06767-1. Epub 2019 Apr 3. PMID 30945059
- [Background] Tighe P, Buckenmaier CC 3rd, Boezaart AP, Carr DB, Clark LL, Herring AA, Kent M, Mackey S, Mariano ER, Polomano RC, Reisfield GM. Acute Pain Medicine in the United States: A Status Report. Pain Med. 2015 Sep;16(9):1806-26. doi: 10.1111/pme.12760. Epub 2015 Jun 10. PMID 26535424
- [Background] Howard R, Fry B, Gunaseelan V, Lee J, Waljee J, Brummett C, Campbell D Jr, Seese E, Englesbe M, Vu J. Association of Opioid Prescribing With Opioid Consumption After Surgery in Michigan. JAMA Surg. 2019 Jan 1;154(1):e184234. doi: 10.1001/jamasurg.2018.4234. Epub 2019 Jan 16. PMID 30422239
- [Background] Ossiander EM. Using textual cause-of-death data to study drug poisoning deaths. Am J Epidemiol. 2014 Apr 1;179(7):884-94. doi: 10.1093/aje/kwt333. Epub 2014 Feb 11. PMID 24521559
- [Background] Banta-Green CJ, Merrill JO, Doyle SR, Boudreau DM, Calsyn DA. Measurement of opioid problems among chronic pain patients in a general medical population. Drug Alcohol Depend. 2009 Sep 1;104(1-2):43-9. doi: 10.1016/j.drugalcdep.2009.03.022. Epub 2009 May 26. PMID 19473787
- [Background] Jones CM, Paulozzi LJ, Mack KA. Sources of prescription opioid pain relievers by frequency of past-year nonmedical use United States, 2008-2011. JAMA Intern Med. 2014 May;174(5):802-3. doi: 10.1001/jamainternmed.2013.12809. No abstract available. PMID 24589763
- [Background] Hill MV, McMahon ML, Stucke RS, Barth RJ Jr. Wide Variation and Excessive Dosage of Opioid Prescriptions for Common General Surgical Procedures. Ann Surg. 2017 Apr;265(4):709-714. doi: 10.1097/SLA.0000000000001993. PMID 27631771
- [Background] Bartels K, Binswanger IA, Hopfer CJ. Sources of Prescription Opioids for Nonmedical Use. J Addict Med. 2016 Mar-Apr;10(2):134. doi: 10.1097/ADM.0000000000000192. No abstract available. PMID 26985647
- [Background] Compton WM, Volkow ND. Major increases in opioid analgesic abuse in the United States: concerns and strategies. Drug Alcohol Depend. 2006 Feb 1;81(2):103-7. doi: 10.1016/j.drugalcdep.2005.05.009. Epub 2005 Jul 14. PMID 16023304
- [Background] Harris K, Curtis J, Larsen B, Calder S, Duffy K, Bowen G, Hadley M, Tristani-Firouzi P. Opioid pain medication use after dermatologic surgery: a prospective observational study of 212 dermatologic surgery patients. JAMA Dermatol. 2013 Mar;149(3):317-21. doi: 10.1001/jamadermatol.2013.1871. PMID 23682368
- [Background] Bates C, Laciak R, Southwick A, Bishoff J. Overprescription of postoperative narcotics: a look at postoperative pain medication delivery, consumption and disposal in urological practice. J Urol. 2011 Feb;185(2):551-5. doi: 10.1016/j.juro.2010.09.088. Epub 2010 Dec 18. PMID 21168869
- [Background] Lankenau SE, Teti M, Silva K, Jackson Bloom J, Harocopos A, Treese M. Initiation into prescription opioid misuse amongst young injection drug users. Int J Drug Policy. 2012 Jan;23(1):37-44. doi: 10.1016/j.drugpo.2011.05.014. Epub 2011 Jun 20. PMID 21689917
- [Background] Inciardi JA, Surratt HL, Cicero TJ, Beard RA. Prescription opioid abuse and diversion in an urban community: the results of an ultrarapid assessment. Pain Med. 2009 Apr;10(3):537-48. doi: 10.1111/j.1526-4637.2009.00603.x. PMID 19416440
- [Background] Volkow ND, McLellan TA. Curtailing diversion and abuse of opioid analgesics without jeopardizing pain treatment. JAMA. 2011 Apr 6;305(13):1346-7. doi: 10.1001/jama.2011.369. No abstract available. PMID 21467287
- [Background] Hill MV, Stucke RS, Billmeier SE, Kelly JL, Barth RJ Jr. Guideline for Discharge Opioid Prescriptions after Inpatient General Surgical Procedures. J Am Coll Surg. 2018 Jun;226(6):996-1003. doi: 10.1016/j.jamcollsurg.2017.10.012. Epub 2017 Nov 30. PMID 29198638
- [Background] Overton HN, Hanna MN, Bruhn WE, Hutfless S, Bicket MC, Makary MA; Opioids After Surgery Workgroup. Opioid-Prescribing Guidelines for Common Surgical Procedures: An Expert Panel Consensus. J Am Coll Surg. 2018 Oct;227(4):411-418. doi: 10.1016/j.jamcollsurg.2018.07.659. Epub 2018 Aug 14. PMID 30118896
- [Background] Glod SA. The Other Victims of the Opioid Epidemic. N Engl J Med. 2017 Jun 1;376(22):2101-2102. doi: 10.1056/NEJMp1702188. No abstract available. PMID 28564563
- [Background] Nair BG, Newman SF, Peterson GN, Wu WY, Schwid HA. Feedback mechanisms including real-time electronic alerts to achieve near 100% timely prophylactic antibiotic administration in surgical cases. Anesth Analg. 2010 Nov;111(5):1293-300. doi: 10.1213/ANE.0b013e3181f46d89. Epub 2010 Sep 14. PMID 20841414
- [Background] Abrams BA, Murray KA, Mahoney K, Raymond KM, McWilliams SK, Nichols S, Mahmoudi E, Mayes LM, Fernandez-Bustamante A, Mitchell JD, Meguid RA, Zanotti G, Bartels K. Postdischarge Pain Management After Thoracic Surgery: A Patient-Centered Approach. Ann Thorac Surg. 2020 Nov;110(5):1714-1721. doi: 10.1016/j.athoracsur.2020.04.048. Epub 2020 Jun 1. PMID 32497643
- [Background] Derry CJ, Derry S, Moore RA. Single dose oral ibuprofen plus paracetamol (acetaminophen) for acute postoperative pain. Cochrane Database Syst Rev. 2013 Jun 24;2013(6):CD010210. doi: 10.1002/14651858.CD010210.pub2. PMID 23794268
- [Background] Valentine AR, Carvalho B, Lazo TA, Riley ET. Scheduled acetaminophen with as-needed opioids compared to as-needed acetaminophen plus opioids for post-cesarean pain management. Int J Obstet Anesth. 2015 Aug;24(3):210-6. doi: 10.1016/j.ijoa.2015.03.006. Epub 2015 Mar 23. PMID 25936786
- [Background] Bouwsma EVA, Huirne JAF, van de Ven PM, Vonk Noordegraaf A, Schaafsma FG, Schraffordt Koops SE, van Kesteren PJM, Brolmann HAM, Anema JR. Effectiveness of an internet-based perioperative care programme to enhance postoperative recovery in gynaecological patients: cluster controlled trial with randomised stepped-wedge implementation. BMJ Open. 2018 Jan 30;8(1):e017781. doi: 10.1136/bmjopen-2017-017781. PMID 29382673
- [Background] Horstman MJ, Mills WL, Herman LI, Cai C, Shelton G, Qdaisat T, Berger DH, Naik AD. Patient experience with discharge instructions in postdischarge recovery: a qualitative study. BMJ Open. 2017 Feb 22;7(2):e014842. doi: 10.1136/bmjopen-2016-014842. PMID 28228448
- [Background] Sanders GD, Neumann PJ, Basu A, Brock DW, Feeny D, Krahn M, Kuntz KM, Meltzer DO, Owens DK, Prosser LA, Salomon JA, Sculpher MJ, Trikalinos TA, Russell LB, Siegel JE, Ganiats TG. Recommendations for Conduct, Methodological Practices, and Reporting of Cost-effectiveness Analyses: Second Panel on Cost-Effectiveness in Health and Medicine. JAMA. 2016 Sep 13;316(10):1093-103. doi: 10.1001/jama.2016.12195. PMID 27623463
- [Background] Stacey D, Bennett CL, Barry MJ, Col NF, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Legare F, Thomson R. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD001431. doi: 10.1002/14651858.CD001431.pub3. PMID 21975733
- [Background] Shojania KG, Jennings A, Mayhew A, Ramsay CR, Eccles MP, Grimshaw J. The effects of on-screen, point of care computer reminders on processes and outcomes of care. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD001096. doi: 10.1002/14651858.CD001096.pub2. PMID 19588323
- [Background] Reilly BM, Evans AT. Translating clinical research into clinical practice: impact of using prediction rules to make decisions. Ann Intern Med. 2006 Feb 7;144(3):201-9. doi: 10.7326/0003-4819-144-3-200602070-00009. PMID 16461965
- [Background] Moons KG, Royston P, Vergouwe Y, Grobbee DE, Altman DG. Prognosis and prognostic research: what, why, and how? BMJ. 2009 Feb 23;338:b375. doi: 10.1136/bmj.b375. No abstract available. PMID 19237405
- [Background] Kansagara D, Englander H, Salanitro A, Kagen D, Theobald C, Freeman M, Kripalani S. Risk prediction models for hospital readmission: a systematic review. JAMA. 2011 Oct 19;306(15):1688-98. doi: 10.1001/jama.2011.1515. PMID 22009101
- [Background] Justice AC, Covinsky KE, Berlin JA. Assessing the generalizability of prognostic information. Ann Intern Med. 1999 Mar 16;130(6):515-24. doi: 10.7326/0003-4819-130-6-199903160-00016. PMID 10075620
- [Background] Moons KG, Altman DG, Vergouwe Y, Royston P. Prognosis and prognostic research: application and impact of prognostic models in clinical practice. BMJ. 2009 Jun 4;338:b606. doi: 10.1136/bmj.b606. No abstract available. PMID 19502216
- [Background] Ryan R, Santesso N, Hill S, Lowe D, Kaufman C, Grimshaw J. Consumer-oriented interventions for evidence-based prescribing and medicines use: an overview of systematic reviews. Cochrane Database Syst Rev. 2011 May 11;(5):CD007768. doi: 10.1002/14651858.CD007768.pub2. PMID 21563160
- [Background] Sessler DI, Myles PS. Novel Clinical Trial Designs to Improve the Efficiency of Research. Anesthesiology. 2020 Jan;132(1):69-81. doi: 10.1097/ALN.0000000000002989. PMID 31809323
- [Background] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159
- [Background] Thorpe KE, Zwarenstein M, Oxman AD, Treweek S, Furberg CD, Altman DG, Tunis S, Bergel E, Harvey I, Magid DJ, Chalkidou K. A pragmatic-explanatory continuum indicator summary (PRECIS): a tool to help trial designers. J Clin Epidemiol. 2009 May;62(5):464-75. doi: 10.1016/j.jclinepi.2008.12.011. PMID 19348971
- [Background] Fernandez-Bustamante A, Bartels K, Clavijo C, Scott BK, Kacmar R, Bullard K, Moss AFD, Henderson W, Juarez-Colunga E, Jameson L. Preoperatively Screened Obstructive Sleep Apnea Is Associated With Worse Postoperative Outcomes Than Previously Diagnosed Obstructive Sleep Apnea. Anesth Analg. 2017 Aug;125(2):593-602. doi: 10.1213/ANE.0000000000002241. PMID 28682951
- [Background] Krause M, McWilliams SK, Bullard KJ, Mayes LM, Jameson LC, Mikulich-Gilbertson SK, Fernandez-Bustamante A, Bartels K. Neostigmine Versus Sugammadex for Reversal of Neuromuscular Blockade and Effects on Reintubation for Respiratory Failure or Newly Initiated Noninvasive Ventilation: An Interrupted Time Series Design. Anesth Analg. 2020 Jul;131(1):141-151. doi: 10.1213/ANE.0000000000004505. PMID 31702700
- [Background] Fernandez-Bustamante A, Frendl G, Sprung J, Kor DJ, Subramaniam B, Martinez Ruiz R, Lee JW, Henderson WG, Moss A, Mehdiratta N, Colwell MM, Bartels K, Kolodzie K, Giquel J, Vidal Melo MF. Postoperative Pulmonary Complications, Early Mortality, and Hospital Stay Following Noncardiothoracic Surgery: A Multicenter Study by the Perioperative Research Network Investigators. JAMA Surg. 2017 Feb 1;152(2):157-166. doi: 10.1001/jamasurg.2016.4065. PMID 27829093
- [Background] Bartels K, Fernandez-Bustamante A, McWilliams SK, Hopfer CJ, Mikulich-Gilbertson SK. Long-term opioid use after inpatient surgery - A retrospective cohort study. Drug Alcohol Depend. 2018 Jun 1;187:61-65. doi: 10.1016/j.drugalcdep.2018.02.013. Epub 2018 Mar 27. PMID 29627407
- [Background] Bartels K, Kaizer A, Jameson L, Bullard K, Dingmann C, Fernandez-Bustamante A. Hypoxemia Within the First 3 Postoperative Days Is Associated With Increased 1-Year Postoperative Mortality After Adjusting for Perioperative Opioids and Other Confounders. Anesth Analg. 2020 Aug;131(2):555-563. doi: 10.1213/ANE.0000000000004553. PMID 31971921
- [Background] Bookman K, West D, Ginde A, Wiler J, McIntyre R, Hammes A, Carlson N, Steinbruner D, Solley M, Zane R. Embedded Clinical Decision Support in Electronic Health Record Decreases Use of High-cost Imaging in the Emergency Department: EmbED study. Acad Emerg Med. 2017 Jul;24(7):839-845. doi: 10.1111/acem.13195. Epub 2017 May 11. PMID 28391603
- [Background] Wellek S, Blettner M. On the proper use of the crossover design in clinical trials: part 18 of a series on evaluation of scientific publications. Dtsch Arztebl Int. 2012 Apr;109(15):276-81. doi: 10.3238/arztebl.2012.0276. Epub 2012 Apr 13. PMID 22567063
- [Background] Turner RM, White IR, Croudace T; PIP Study Group. Analysis of cluster randomized cross-over trial data: a comparison of methods. Stat Med. 2007 Jan 30;26(2):274-89. doi: 10.1002/sim.2537. PMID 16538700
- [Background] Reich NG, Myers JA, Obeng D, Milstone AM, Perl TM. Empirical power and sample size calculations for cluster-randomized and cluster-randomized crossover studies. PLoS One. 2012;7(4):e35564. doi: 10.1371/journal.pone.0035564. Epub 2012 Apr 27. PMID 22558168
- [Background] Arnup SJ, McKenzie JE, Hemming K, Pilcher D, Forbes AB. Understanding the cluster randomised crossover design: a graphical illustraton of the components of variation and a sample size tutorial. Trials. 2017 Aug 15;18(1):381. doi: 10.1186/s13063-017-2113-2. PMID 28810895
- [Background] Murray DM, Varnell SP, Blitstein JL. Design and analysis of group-randomized trials: a review of recent methodological developments. Am J Public Health. 2004 Mar;94(3):423-32. doi: 10.2105/ajph.94.3.423. PMID 14998806
- [Background] Milani RV, Franklin NC. The Role of Technology in Healthy Living Medicine. Prog Cardiovasc Dis. 2017 Mar-Apr;59(5):487-491. doi: 10.1016/j.pcad.2017.02.001. Epub 2017 Feb 11. PMID 28189614
- [Background] Krebs P, Duncan DT. Health App Use Among US Mobile Phone Owners: A National Survey. JMIR Mhealth Uhealth. 2015 Nov 4;3(4):e101. doi: 10.2196/mhealth.4924. PMID 26537656
- [Background] Liu VX, Rosas E, Hwang J, Cain E, Foss-Durant A, Clopp M, Huang M, Lee DC, Mustille A, Kipnis P, Parodi S. Enhanced Recovery After Surgery Program Implementation in 2 Surgical Populations in an Integrated Health Care Delivery System. JAMA Surg. 2017 Jul 19;152(7):e171032. doi: 10.1001/jamasurg.2017.1032. Epub 2017 Jul 19. PMID 28492816
- [Background] Tobias JD, Green TP, Cote CJ; SECTION ON ANESTHESIOLOGY AND PAIN MEDICINE; COMMITTEE ON DRUGS. Codeine: Time to Say "No". Pediatrics. 2016 Oct;138(4):e20162396. doi: 10.1542/peds.2016-2396. Epub 2016 Sep 19. PMID 27647717
- [Background] Barozzi N, Tett SE. Perceived barriers to paracetamol (acetaminophen) prescribing, especially following rofecoxib withdrawal from the market. Clin Rheumatol. 2009 May;28(5):509-19. doi: 10.1007/s10067-008-1077-8. Epub 2009 Jan 9. PMID 19132456
- [Background] Sirey JA, Banerjee S, Marino P, Bruce ML, Halkett A, Turnwald M, Chiang C, Liles B, Artis A, Blow F, Kales HC. Adherence to Depression Treatment in Primary Care: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Nov 1;74(11):1129-1135. doi: 10.1001/jamapsychiatry.2017.3047. PMID 28973066
- [Background] Campbell AN, Nunes EV, Matthews AG, Stitzer M, Miele GM, Polsky D, Turrigiano E, Walters S, McClure EA, Kyle TL, Wahle A, Van Veldhuisen P, Goldman B, Babcock D, Stabile PQ, Winhusen T, Ghitza UE. Internet-delivered treatment for substance abuse: a multisite randomized controlled trial. Am J Psychiatry. 2014 Jun;171(6):683-90. doi: 10.1176/appi.ajp.2014.13081055. PMID 24700332
- [Background] Dong Y, Wang P, Dai Z, Liu K, Jin Y, Li A, Wang S, Zheng J. Increased self-care activities and glycemic control rate in relation to health education via Wechat among diabetes patients: A randomized clinical trial. Medicine (Baltimore). 2018 Dec;97(50):e13632. doi: 10.1097/MD.0000000000013632. PMID 30558051
- [Background] Attum B, Rodriguez-Buitrago A, Harrison N, Evans A, Obremskey W, Sethi MK, Jahangir AA. Opioid Prescribing Practices by Orthopaedic Trauma Surgeons After Isolated Femur Fractures. J Orthop Trauma. 2018 Mar;32(3):e106-e111. doi: 10.1097/BOT.0000000000001046. PMID 29065039
- [Background] Dhumane PW, Diana M, Leroy J, Marescaux J. Minimally invasive single-site surgery for the digestive system: A technological review. J Minim Access Surg. 2011 Jan;7(1):40-51. doi: 10.4103/0972-9941.72381. PMID 21197242
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Ellis TD, Cavanaugh JT, DeAngelis T, Hendron K, Thomas CA, Saint-Hilaire M, Pencina K, Latham NK. Comparative Effectiveness of mHealth-Supported Exercise Compared With Exercise Alone for People With Parkinson Disease: Randomized Controlled Pilot Study. Phys Ther. 2019 Feb 1;99(2):203-216. doi: 10.1093/ptj/pzy131. PMID 30715489
- [Background] White IR, Horton NJ, Carpenter J, Pocock SJ. Strategy for intention to treat analysis in randomised trials with missing outcome data. BMJ. 2011 Feb 7;342:d40. doi: 10.1136/bmj.d40. PMID 21300711
- [Background] Brainard J, Scott BK, Sullivan BL, Fernandez-Bustamante A, Piccoli JR, Gebbink MG, Bartels K. Heated humidified high-flow nasal cannula oxygen after thoracic surgery - A randomized prospective clinical pilot trial. J Crit Care. 2017 Aug;40:225-228. doi: 10.1016/j.jcrc.2017.04.023. Epub 2017 Apr 19. PMID 28454060
- [Background] Teja BJ, Sutherland TN, Barnett SR, Talmor DS. Cost-Effectiveness Research in Anesthesiology. Anesth Analg. 2018 Nov;127(5):1196-1201. doi: 10.1213/ANE.0000000000003334. PMID 29570150
- [Background] Carias C, Chesson HW, Grosse SD, Li R, Meltzer MI, Miller GF, Murphy LB, Nurmagambetov TA, Pike JJ, Whitham HK. Recommendations of the Second Panel on Cost Effectiveness in Health and Medicine: A Reference, Not a Rule Book. Am J Prev Med. 2018 Apr;54(4):600-602. doi: 10.1016/j.amepre.2017.11.013. Epub 2018 Jan 12. No abstract available. PMID 29338958
- [Background] Wang H, Li T, Siahpush M, Chen LW, Huberty J. Cost-Effectiveness of Ready for Recess to Promote Physical Activity in Children. J Sch Health. 2017 Apr;87(4):278-285. doi: 10.1111/josh.12495. PMID 28260240
- [Background] Neary KC, Mormino MA, Wang H. Suture Button Fixation Versus Syndesmotic Screws in Supination-External Rotation Type 4 Injuries: A Cost-Effectiveness Analysis. Am J Sports Med. 2017 Jan;45(1):210-217. doi: 10.1177/0363546516664713. Epub 2016 Sep 30. PMID 27601151
- [Background] Grimsrud C, Killen C, Murphy M, Wang H, McGarry S. Long-Term Outcomes of Rotationplasty patients in the treatment of lower extremity sarcomas with cost analysis. J Clin Orthop Trauma. 2020 Feb;11(Suppl 1):S149-S152. doi: 10.1016/j.jcot.2019.06.003. Epub 2019 Jun 5. PMID 31992936
- [Background] Young L, Zimmerman L, Pozehl B, Barnason S, Wang H. Cost-effectiveness of a symptom management intervention: improving physical activity in older women following coronary artery bypass surgery. Nurs Econ. 2012 Mar-Apr;30(2):94-103. PMID 22558727
- [Background] Wang H, Qiu F, Boilesen E, Nayar P, Lander L, Watkins K, Watanabe-Galloway S. Rural-Urban Differences in Costs of End-of-Life Care for Elderly Cancer Patients in the United States. J Rural Health. 2016 Sep;32(4):353-362. doi: 10.1111/jrh.12160. Epub 2015 Nov 20. PMID 26586101
- [Background] Wang H, Gregg A, Qiu F, Kim J, Chen B, Wan N, Su D, Michaud T, Chen LW. Breast Cancer Screening for Patients of Rural Accountable Care Organization Clinics: A Multi-Level Analysis of Barriers and Facilitators. J Community Health. 2018 Apr;43(2):248-258. doi: 10.1007/s10900-017-0412-x. PMID 28861654
- [Background] McClure NS, Sayah FA, Xie F, Luo N, Johnson JA. Instrument-Defined Estimates of the Minimally Important Difference for EQ-5D-5L Index Scores. Value Health. 2017 Apr;20(4):644-650. doi: 10.1016/j.jval.2016.11.015. Epub 2017 Jan 10. PMID 28408007
- [Background] Pickard AS, Law EH, Jiang R, Pullenayegum E, Shaw JW, Xie F, Oppe M, Boye KS, Chapman RH, Gong CL, Balch A, Busschbach JJV. United States Valuation of EQ-5D-5L Health States Using an International Protocol. Value Health. 2019 Aug;22(8):931-941. doi: 10.1016/j.jval.2019.02.009. Epub 2019 May 25. PMID 31426935
- [Background] Shaw JW, Johnson JA, Coons SJ. US valuation of the EQ-5D health states: development and testing of the D1 valuation model. Med Care. 2005 Mar;43(3):203-20. doi: 10.1097/00005650-200503000-00003. PMID 15725977
- [Background] Schwarzer R, Rochau U, Saverno K, Jahn B, Bornschein B, Muehlberger N, Flatscher-Thoeni M, Schnell-Inderst P, Sroczynski G, Lackner M, Schall I, Hebborn A, Pugner K, Fehervary A, Brixner D, Siebert U. Systematic overview of cost-effectiveness thresholds in ten countries across four continents. J Comp Eff Res. 2015 Sep;4(5):485-504. doi: 10.2217/cer.15.38. PMID 26490020
- [Background] Claxton K, Sculpher M, McCabe C, Briggs A, Akehurst R, Buxton M, Brazier J, O'Hagan T. Probabilistic sensitivity analysis for NICE technology assessment: not an optional extra. Health Econ. 2005 Apr;14(4):339-47. doi: 10.1002/hec.985. PMID 15736142
- [Background] Cantor SB. Cost-effectiveness analysis, extended dominance, and ethics: a quantitative assessment. Med Decis Making. 1994 Jul-Sep;14(3):259-65. doi: 10.1177/0272989X9401400308. PMID 7934713
- [Derived] Rolfzen ML, Shah K, Sanchez Rodriguez E, Hoffman JT, Clauw D, Mascha E, Graff V, Bartels K. Postsurgical Medication Awareness, Recovery, and Tracking using a Phone-Based App (SMART-APP): a randomized clinical trial. Reg Anesth Pain Med. 2025 Jul 2:rapm-2025-106783. doi: 10.1136/rapm-2025-106783. Online ahead of print. PMID 40602806

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from May 2, 2022 to December 10, 2023. Participants were enrolled in the hospital setting.
Groups:
- UControlPain App With Only Data Collection: UControlPain App with only data collection function. No provider-facing tool.
- UControlPain Educational App: UControlPain app with education components. No provider-facing tool.
- UControlPain App and Provider Facing Tool: UControlPain app with education components and provider-facing prescription intervention. Participants who were randomized to the intervention arm (UControlPain App) once half the subjects were enrolled (February 13, 2023).
- UControlPain App With Only Data Collection and Provider Facing Tool: UControlPain App with only data collection function and Provider-facing prescription intervention. Participants who were randomized to the control arm (UControlPain App with only data collection), once half the subjects were enrolled (February 13, 2023).
Period: Overall Study
Arm/Group | UControlPain App With Only Data Collection | UControlPain Educational App | UControlPain App and Provider Facing Tool | UControlPain App With Only Data Collection and Provider Facing Tool
Started | 179 | 179 | 176 | 177
Completed | 152 | 148 | 155 | 151
Not Completed | 27 | 31 | 21 | 26
Not completed — Withdrawal by Subject | 5 | 7 | 6 | 4
Not completed — Physician Decision | 3 | 2 | 1 | 4
Not completed — Lost to Follow-up | 12 | 17 | 14 | 14
Not completed — Discharge plan revised; app compatibility issue or chronic opioid use discovered post-enrollment. | 7 | 5 | 0 | 4

BASELINE CHARACTERISTICS:
Population: A total of 711 participants consented to the trial, and 606 completed the research.
Groups:
- UControlPain App With Only Data Collection Function: UControlPain App with only data collection function. No provider-facing tool.
- UControlPain Educational App Only: UControl Pain App with education components only. No provider-facing tool.
- Total: Total of all reporting groups
Arm/Group | UControlPain App With Only Data Collection Function | UControlPain Educational App Only | UControlPain App and Provider Facing Tool | UControlPain App With Only Data Collection and Provider Facing Tool | Total
Number analyzed (Participants) | 179 | 179 | 176 | 177 | 711
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 154 | 145 | 146 | 150 | 595
  >=65 years | 25 | 34 | 30 | 27 | 116
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 108 | 110 | 123 | 455
  Male | 65 | 71 | 66 | 54 | 256
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 9 | 12 | 36
  Not Hispanic or Latino | 170 | 171 | 167 | 165 | 673
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 2 | 0 | 5
  Asian | 1 | 1 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 15 | 11 | 20 | 13 | 59
  White | 154 | 155 | 145 | 151 | 605
  More than one race | 0 | 2 | 3 | 1 | 6
  Unknown or Not Reported | 8 | 7 | 4 | 10 | 29
Region of Enrollment [Number; unit: participants]
  United States | 179 | 179 | 176 | 177 | 711

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Weekly Opioid Intake After Discharge
Description: Opioids reported as taken will be recorded by type of opioid, units, and total amount taken within the first 28 days after hospital discharge. To account for different opioid potencies, the cumulative dose of opioids will be expressed in milligram morphine equivalents (MME).
Time Frame: Baseline (discharge), weekly for four weeks
Population: Participants who completed at least one week of surveys were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Morphine milligram equivalents
Groups:
- UControlPain Educational App: UControl Pain App with education components only. No provider-facing tool.
Arm/Group | UControlPain Educational App | UControlPain App With Only Data Collection | UControlPain App and Provider Facing Tool | UControlPain App With Only Data Collection and Provider Facing Tool
Number analyzed (Participants) | 148 | 152 | 155 | 151
Morphine milligram equivalents | 30 [0 to 105] | 30 [0 to 76.9] | 20 [0 to 90] | 10 [0 to 81.8]

2. Secondary Outcome: Pain Assessment-Pain Intensity
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) was used to measure pain intensity, with higher scores indicating more intense pain. The PROMIS was assessed four times after discharge, once per week for 28 days, and averaged. On the PROMIS 4-item scale pain intensity scores, higher scores indicate higher pain intensity. All PROMIS scores are analyzed as standardized T-scores [mean=50, standard deviation (SD) =10].
Time Frame: Weekly for four weeks after discharge
Population: Subjects who completed at least one week of surveys were included in the analysis.
Measure: Median (Standard Deviation); unit: T-score
Groups:
- UControlPain Educational App: UControl Pain App with education components. No provider-facing tool.
- UControlPain App With Only Data Collection: Control UControl Pain App with data collection only. No provider-facing tool.
Arm/Group | UControlPain Educational App | UControlPain App With Only Data Collection | UControlPain App and Provider Facing Tool | UControlPain App With Only Data Collection and Provider Facing Tool
Number analyzed (Participants) | 148 | 152 | 155 | 151
T-score | 52.5 (9.89) | 51.24 (9.37) | 52.51 (9.48) | 51.29 (9.06)

3. Secondary Outcome: Pain Assessment-Pain Interference
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) was used to measure pain interference, with higher scores indicating more intense pain. The PROMIS was assessed four times after discharge, once per week for 28 days, and averaged. On the PROMIS 4-item scale pain interference scores, higher scores indicate higher pain interference. All PROMIS scores are analyzed as standardized T-scores [mean=50, standard deviation (SD) =10].
Time Frame: Weekly for four weeks after discharge
Population: Subjects who completed at least one week of surveys were included in the analysis.
Measure: Median (Standard Deviation); unit: T-score
Arm/Group | UControlPain Educational App | UControlPain App With Only Data Collection | UControlPain App and Provider Facing Tool | UControlPain App With Only Data Collection and Provider Facing Tool
Number analyzed (Participants) | 148 | 152 | 155 | 151
T-score | 55.28 (9.79) | 54.17 (9.95) | 55.13 (9.34) | 53.43 (9.62)

4. Secondary Outcome: Opioid Prescription Amount in Morphine Milligram Equivalents on Day of Discharge
Description: Opioids prescribed on the day of discharge will be recorded by type of opioid, unit dispensed, and total amount dispensed. To account for different opioid potencies, the cumulative dose of opioids will be expressed in milligram morphine equivalents (MME).
Time Frame: Baseline (discharge)
Population: Subjects who completed at least one week of surveys were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: Morphine milligram equivalents
Arm/Group | UControlPain Educational App | UControlPain App With Only Data Collection | UControlPain App and Provider Facing Tool | UControlPain App With Only Data Collection and Provider Facing Tool
Number analyzed (Participants) | 148 | 152 | 155 | 151
Morphine milligram equivalents | 90 [60 to 150] | 77.5 [60 to 157.5] | 75.0 [56.2 to 150.0] | 75.0 [40 to 150]

5. Secondary Outcome: Number of Participants With Opioids Prescribed From "Day of Discharge + 1" Until 28 Days After Discharge
Description: Discovered by medical record review. This measure will account for opioids prescribed to patients because they run out prematurely. We will calculate opioid prescriptions from "day of discharge +1" until 28 days after discharge.
Time Frame: Baseline (discharge) +1 day until day 28, up to 27 days total
Population: Subjects who completed at least one week of surveys were included in the data analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | UControlPain Educational App | UControlPain App With Only Data Collection | UControlPain App and Provider Facing Tool | UControlPain App With Only Data Collection and Provider Facing Tool
Number analyzed (Participants) | 148 | 152 | 155 | 151
Participants | 23 | 21 | 31 | 25

6. Secondary Outcome: Number of Participants Who Disposed of Opioids
Description: Number of participants who reported their disposal of any leftover opioids is recorded. This is reported on the weekly surveys done in 28 days post-discharge.
Time Frame: Baseline (discharge), weekly for four weeks
Population: Participants who answered they had opioids left over were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | UControlPain Educational App | UControlPain App With Only Data Collection | UControlPain App and Provider Facing Tool | UControlPain App With Only Data Collection and Provider Facing Tool
Number analyzed (Participants) | 148 | 152 | 155 | 151
Participants | 3 | 2 | 3 | 6

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Discharge to Day 28.
Description: 1. All-Cause Mortality: all anticipated and unanticipated deaths due to any cause.
  2. Serious Adverse Events: all anticipated and unanticipated serious adverse events, including only inpatient hospitalization
  3. Other (Not Including Serious) Adverse Events: A table of anticipated and unanticipated events
Groups:
- UControl Pain App Educational App: UControl Pain App with education components. No provider-facing tool.
Arm/Group | UControl Pain App Educational App | UControlPain App With Only Data Collection | UControlPain App and Provider Facing Tool | UControlPain App With Only Data Collection and Provider Facing Tool
All-Cause Mortality (participants affected / at risk) | 0/148 | 1/152 | 0/155 | 0/151
Serious Adverse Events (participants affected / at risk) | 11/148 | 12/152 | 8/155 | 11/151
Other Adverse Events (participants affected / at risk) | 2/148 | 1/152 | 0/155 | 0/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UControl Pain App Educational App (N=148) | UControlPain App With Only Data Collection (N=152) | UControlPain App and Provider Facing Tool (N=155) | UControlPain App With Only Data Collection and Provider Facing Tool (N=151)
Re-hospitalization (any reason) (Surgical and medical procedures) | 11 (11) | 12 (12) | 8 (8) | 11 (11)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UControl Pain App Educational App (N=148) | UControlPain App With Only Data Collection (N=152) | UControlPain App and Provider Facing Tool (N=155) | UControlPain App With Only Data Collection and Provider Facing Tool (N=151)
Requiring greater than 2 additional opioid prescriptions within 2 weeks of discharge (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT05221866/Prot_SAP_002.pdf
  • Informed Consent Form (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT05221866/ICF_003.pdf